CLINICAL TRIAL: NCT04277546
Title: A Phase 2 Open-label, Long-term Extension Safety Study of Brazikumab in Participants With Moderately to Severely Active Ulcerative Colitis (EXPEDITION OLE)
Brief Title: Open-label Extension Study of Brazikumab in Ulcerative Colitis
Acronym: Expedition
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision to discontinue the development of brazikumab in inflammatory bowel disease.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5272C00002; #3151-202-008 (Other: Legacy); 2021-001644-10 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brazikumab Maintenance Dose (Experimental): Administer at 4-week intervals through Week 52 Participants who receive IV induction dosing will be administered brazikumab SC at 4-week intervals starting Week 12 through Week 52
  Interventions: Drug: Brazikumab Maintenance Dose
- Brazikumab Induction Dose (Experimental): Administer at Week 0, Week 4, and Week 8
  Interventions: Drug: Brazikumab Induction Dose

INTERVENTIONS:
Drug: Brazikumab Maintenance Dose — Completers in the lead-in study D5272C00001 (Legacy #3151-201-008) will receive a maintenance dose of brazikumab administered subcutaneously every 4 weeks up to Week 52 (Group A). The SC dose of brazikumab will be administered to all responders/completers in the lead-in study regardless of the prior treatment administered.
  Arms: Brazikumab Maintenance Dose
Drug: Brazikumab Induction Dose — Participants in the lead-in study D5272C00001 (Legacy #3151-201-008) who have not responded to treatment and have met criteria for rescue treatment are considered inadequate/non-responders (Group B). In these eligible participants, IV induction dosing of brazikumab at Week 0, Week 4, and Week 8 will be administered, followed by brazikumab administered subcutaneously every 4 weeks thereafter (up to Week 52).
  Arms: Brazikumab Induction Dose

SUMMARY:
The purpose of this OLE Study D5272C00002 (Legacy #3151-202-008) is to permit participants who previously enrolled in the double-blind Study D5272C00001 (Legacy #3151-201-008) to receive brazikumab, allowing for long-term observation of safety and efficacy in these participants treated with brazikumab. There are no formal hypotheses to be tested. Safety and efficacy data obtained in this study will be included in regulatory product submissions as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1.01 Male or female participants who: successfully completed or discontinued participation due to lack of efficacy after Week 10 in the lead-in Study D5272C00001 (Legacy #3151-201-008). AND Meets 1 of the following criteria for successful completion or early termination from Study D5272C00001 (Legacy #3151-201-008):

1. Participant completed Study D5272C00001 (Legacy #3151-201-008), received scheduled study interventions, completed scheduled visits, and completed Week 54 assessments.
2. Participant discontinued participation due to lack of efficacy after Week 10 in Study D5272C00001 (Legacy #3151-201-008), received scheduled study interventions, and completed Early Termination Visit assessments.

1.02. Deleted Eligibility as part of Amendment 2 1.03. Deleted Eligibility as part of Amendment 3 1.04. Deleted eligibility as part of Amendment 2 2.01. Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. Nonsterilized men who are sexually active with a female partner of childbearing potential should use condom during treatment and for 18 weeks after the last dose of study intervention, must comply with the methods of contraception described in Criterion 2.02 below, and must not donate or bank sperm for fertilization purpose for the same time period.

2.02. Female participants of childbearing potential must have a negative urine pregnancy test prior to administration of study intervention and must agree to use a highly effective method of birth control (confirmed by the investigator) from signing the ICF throughout the study duration and for at least 18 weeks after last dose of study intervention 2.03. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal.

3.01. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Written informed consent from the participant has been obtained prior to any study related procedures.

Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information [US sites] and written Data Protection consent [EU sites]).

4.01. Demonstration of adequate compliance with the study procedures in Study D5272C00001 (Legacy #3151-201-008), in the opinion of the investigator and/or sponsor.

4.02. Willingness and ability to attend all study visits, comply with the study procedures, and be able to complete the study period.

5.01 Participant must be 18 to 80 years of age inclusive, at the time of signing the ICF.

Complete inclusion criteria are in the study protocol

Exclusion Criteria:

1.01. Any participant with an unresolved AE from the lead-in study that, in the investigator's opinion, would limit the participant's ability to participate in or complete this study. Any unresolved AE related to an infection will require further discussion with the study physician/designee prior to enrollment.

1.02. Current diagnosis of fulminant colitis, CD or indeterminate colitis, presence of a fistula consistent with CD, primary sclerosing cholangitis, celiac disease, or toxic megacolon. Bile acid malabsorption and other conditions that may potentially confound assessments must be treated prior to baseline.

1.03. Organ or cell-based transplantation with the exception of corneal transplant.

1.04. Any other condition or finding that, in the investigator's or sponsor's opinion, would either confound proper interpretation of the study or expose a participant to unacceptable risk.

1.05. The following are exclusionary with regards to malignancy:

1. Evidence of intestinal epithelial dysplasia on endoscopy, and this is confirmed on biopsy, the participant must be excluded.
2. Any diagnosis of malignancy that requires discontinuation of study intervention from lead-in study.
3. Any new diagnosis of malignancy after completion of the lead-in study. d) Carcinoma in situ of the cervix, with apparent successful curative therapy within 12 months prior to Week 0.

1.06. Participant meets criteria for discontinuation of study intervention during prior lead-in study.

1.07. Deleted exclusion criterion as part of Amendment 3 1.08. Known history of primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection, including HIV infection.

1.09. Prolonged QTcF interval or conditions leading to additional risk for QT prolongation. Participants with electrolyte abnormalities such as hypokalemia and hypomagnesemia that would increase the risk of QT prolongation are to be corrected prior to enrollment.

1.010. Clinically significant kidney disease including but not limited to:

(a) Chronic kidney disease with an estimated glomerular filtration rate of less than 30 ml/min calculated by Modification of Diet in Renal Disease equation, asapplicable, by the central laboratory at screening are excluded.

2.01. Participant requires additional immunosuppressive therapy (aside from permitted concomitant medication in the protocol), biological treatment or prohibited treatment 2.02. Deleted eligibility as part of Amendment 2 2.03. Participant received a prohibited medication during participation in the D5272C00001 (Legacy #3151-201-008) study.

2.04. Participant received a Bacille Calmette-Guérin vaccination within 12 months of Week 0 or any other live vaccine < 4 weeks prior to Week 0, or is planning to receive any such vaccine over the course of the study.

2.05. Participant has received an investigational product after discontinuation from Study D5272C00001 (Legacy #3151-201-008) and prior to enrolling in this study or participant is planning to receive an investigational drug (other than study intervention) or investigational device at any time during Study D5272C00002 (Legacy #3151-202-008).

3.01. Participant who discontinued participation due to lack of efficacy after Week 10 in Study D5272C00001 and did not receive all 3 IV infusions of study interventions scheduled for Week 0 (Day 1), Week 2 (Day 15), and Week 6 (Day 43), and SC at Week 10 (Day 71) in accordance with the protocol for Study D5272C00001.

3.02. Participant who discontinued due to lack of efficacy after Week 10 in Study D5272C00001 (Legacy #3151-201-008) but currently demonstrates clinical response and/or meets endoscopic Mayo Score of 0 or 1 prior to Week 54 in Study D5272C00001 (Legacy #3151-201-008): Clinical Response defined as: Reduction in mMS ≥ 2 points from baseline AND ≥ 30% from baseline, AND a decrease in the rectal bleeding score ≥ 1 point from baseline or a score of 0 or 1, in Study D5272C00001 (Legacy #3151-201-008). Note: Participants are encouraged to remain in the lead-in Study D5272C00001 (Legacy #3151-201-008) if the participant is demonstrating evidence of clinical response. Participants should not early terminate that study due to lack of efficacy if this exclusion is met.

4.01. Abnormal laboratory results at screening as described in the protocol. 5.01. Females who are pregnant, breast feeding, or planning a pregnancy during the study OR females who are of childbearing potential and do not agree to use contraception consistently and correctly as required by the study protocol.

5.02. Participant is directly or indirectly involved in the planning and/or conduct and administration of this study as study staff member, or employee of the sponsor, or the participant is a first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or the participant is enrolled in this study at another clinical study site.

5.03. Judgment that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

5.04. Previous enrollment in the present study.

Complete exclusion criteria are in the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with adverse events | Through week 70
  Number and percentage of patients with reported adverse events.
Percentage of patients with potentially clinically significant changes in laboratory values | Through week 70
  Percentage of patients with potentially clinically significant changes in hematology, clinical chemistry, urinalysis.
Percentage of patients with potentially clinically significant changes in vital signs | Through week 70
  Percentage of patients with potentially clinically significant changes in systolic and diastolic blood pressure, and pulse rate.
Percentage of patients with potentially clinically significant changes in physical exams | Through week 70
  Percentage of patients with potentially clinically significant changes in full physical exams.
Percentage of patients with potentially clinically significant changes in ECGs | Through week 70
  Percentage of patients with potentially clinically significant changes in 12-lead ECG recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Bohannon, Study Director — AstraZeneca
Locations (34):
- United States (10):
  - Research Site, Chula Vista, California
  - Research Site, Lancaster, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Evansville, Indiana
  - Research Site, Beachwood, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Humble, Texas
- Czechia (2):
  - Research Site, České Budějovice
  - Research Site, Ostrava
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Ulm
- Israel (2):
  - Research Site, Haifa
  - Research Site, Jerusalem
- Italy (3):
  - Research Site, Milan
  - Research Site, Rho
  - Research Site, Roma
- Japan (3):
  - Research Site, Kasama-shi
  - Research Site, Kashiwa-shi
  - Research Site, Minatoku
- Poland (5):
  - Research Site, Krakow
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Plumstead
- Research Site, Wŏnju, South Korea
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home